CLINICAL TRIAL: NCT07112495
Title: Evaluation of the Effect of Vaginal Delivery With Labor Analgesia on Maternal Burnout, Breastfeeding Self-Efficacy and Attachment Level
Brief Title: Maternal Burnout, Breastfeeding Self-Efficacy and Attachment Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Prof, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OznurT.
Record Dates: First submitted 2025-05-14; First posted 2025-08-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy
Keywords: pregnancy; pain; burnout; breastfeeding
MeSH Terms: conditions — Pain; Burnout, Psychological; Breast Feeding

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): pregnant women receiving epidural
  Interventions: Other: pregnant women with
- Control (No Intervention): no pregnant women receiving epidural

INTERVENTIONS:
Other: pregnant women with — pregnant women with
  Arms: intervention

SUMMARY:
Labor pain causes women to be afraid of vaginal delivery and to be anxious about delivery and therefore to prefer cesarean delivery (Ali Alahmari et al., 2020). The World Health Organization (WHO) has set the safe cesarean section rate for countries at 15% (World Health Organization, 2015). However, many countries are well above this rate (Betran et al., 2021). An important factor in the preference for cesarean deliveries is the fear of vaginal delivery (Zhao et al., 2021). Vaginal delivery with epidural anesthesia in primiparous women is a very good opportunity to prevent the preference of cesarean deliveries due to fear of vaginal delivery. Unless contraindicated, epidural analgesia should be offered to women to alleviate the pain felt with contractions during labor (Callahan et al., 2023).

Recently, women frequently prefer epidural anesthesia to avoid pain during vaginal delivery. Vaginal delivery with epidural anesthesia aims to minimize the pain of women during the trauma process and is the most effective pain method among pharmacological and nonpharmacological interventions (Antonakou, & Papoutsis, 2016). The reason why vaginal delivery with epidural anesthesia is not widespread enough is that women are not given enough information about epidural anesthesia (Shishido et al., 2020).

DETAILED DESCRIPTION:
Purpose: The aim of this study is to emphasize the importance of vaginal birth with epidural anesthesia in primiparous women (who will have their first birth) in order to reduce the effect of fear of vaginal birth on the choice of cesarean section and to evaluate the effect of increasing the level of knowledge about epidural anesthesia on birth preferences.

Objectives:

To determine the level of fear and anxiety of women regarding childbirth.

To examine the effect of fear of vaginal birth on the preference for cesarean section.

To evaluate the effectiveness of vaginal birth with epidural anesthesia in pain management.

To determine the level of knowledge of women about epidural anesthesia.

To increase the rate of preference for vaginal birth by providing information about epidural anesthesia.

To reveal the role of widespread use of epidural anesthesia in reducing cesarean section rates.

ELIGIBILITY:
Inclusion Criteria:

* Having a normal vaginal delivery in the delivery room,
* 19 to 45 years old
* To be transferred to the Puerperium service after delivery,
* The baby's APGAR score is 7 and above
* 37 and above weeks of gestation
* No complications in the baby and mother due to childbirth
* Postnatal care by the mother's side
* Mother and baby sharing the same room after birth until discharge,
* The mother is breastfeeding her baby,
* Mother's voluntary participation in the study.

Exclusion Criteria:

* Separation of mother and baby for any reason while the mother is with the baby
* Transfer of the baby to the NICU
* Wanting to get out of the study.
* Being a single parent
* Those who cannot speak and write Turkish

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women in labor
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
To determine the breastfeeding self-efficacy levels of mothers. | 1 year
  Assessed using the Breastfeeding Self-Efficacy Scale The minimum possible score on the scale is 14, and the maximum is 70. There is no cutoff point for the scale, and a higher score indicates higher breastfeeding self-efficacy.
To evaluate maternal attachment levels. | 1 year
  Measured with a validated maternal attachment scale. The lowest possible score on the scale is 26, and the highest is 104. A higher score indicates a higher level of maternal attachment.
To examine the breastfeeding status of infants during the first six months of life. | 1 year
  Including exclusive breastfeeding, partial breastfeeding, and formula supplementation
To monitor infant growth and development through percentile tracking during the first six months. | 1 year
  Based on weight, height, and head circumference measurements compared with growth charts

CONTACTS AND LOCATIONS:
Overall Officials: Tiryaki, Study Chair — Sakarya
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: DOI: 10.14744/DAJPNS.2023.00212 — https://dusunenadamdergisi.org/article/1609
- See also: Related Info — https://dusunenadamdergisi.org/article/1609